CLINICAL TRIAL: NCT02916446
Title: Safety Study of Viaskin Peanut to Treat Peanut Allergy
Acronym: REALISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REALISE
Expanded Access: NCT04371627 (No longer available)
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Viaskin Peanut 250 mcg (Experimental): Viaskin Peanut 250 mcg, daily administration
  Interventions: Biological: Viaskin Peanut 250 mcg
- Placebo (Placebo Comparator): Placebo patch, daily administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Viaskin Peanut 250 mcg
  Arms: Viaskin Peanut 250 mcg
Biological: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the safety of Viaskin Peanut 250 mcg in the treatment of peanut allergy in children from 4 to 11 years of age. Subjects will receive either Viaskin Peanut 250 mcg or a placebo for a period of 6 months, after which all subjects will be receiving the active treatment up to a period of 3 years under active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed peanut allergy;
* A peanut Skin Prick Test (SPT) with a wheal largest diameter ≥8 mm;
* A specific-peanut Immunoglobulin E (IgE) ≥14 kU/L;
* Subjects following a strict peanut-free diet.

Exclusion Criteria:

* Generalized dermatologic disease
* Spirometry forced expiratory volume in 1 second (FEV1) <80% of the predicted value, or peak expiratory flow (PEF) <80% of predicted value;
* Receiving β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy; anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy;
* Prior or concomitant history of any immunotherapy to any food allergy (for example EPIT, OIT, SLIT, or specific oral tolerance induction).

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 393 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09-22 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs), Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Through study completion, an average of 3 years

OTHER OUTCOMES:
Change in peanut-specific Immunoglobulins E (IgE) | Baseline, month 3, 6, 9, 12, 18, 24, 30, 36, 42
Change in peanut-specific Immunoglobulins G4 (IgG4) | Baseline, month 3, 6, 9, 12, 18, 24, 30, 36, 42

CONTACTS AND LOCATIONS:
Locations (32):
- United States (26):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Palos Verdes Medical Group, Rolling Hills Estates, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Sarasota Clinical Research, Sarasota, Florida
  - Atlanta Allergy & Asthma Clinic, Marietta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of CHicago, Chicago, Illinois
  - Sneeze, Wheeze and Itch Associates,Clinical Research, Normal, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens' Hospital, Boston, Massachusetts
  - Clinical Research Institute, Plymouth, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Asthma and Allergy Center, Bellevue, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - The University of North Carolina - Chapell Hill, Chapel Hill, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research, Charleston, South Carolina
  - Children's Medical Center of Dallas, Dallas, Texas
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - Sylvana Research, San Antonio, Texas
  - STAAMP Research, San Antonio, Texas
  - ASTHMA, Inc. Clinical Research, Seattle, Washington
- Canada (6):
  - Children's and Women's Health Centre of Brisith Columbia, Vancouver, British Columbia
  - Alpha Medical Research Inc., Mississauga, Ontario
  - Ottawa Allergy Asthma Research Institute, Ottawa, Ontario
  - Gordon Sussman Clinical Research Inc., Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec
  - Centre De Recherche Applique, Québec

REFERENCES:
- [Derived] Pongracic JA, Gagnon R, Sussman G, Siri D, Oriel RC, Brown-Whitehorn TF, Anvari S, Berger WE, Bird JA, Chan ES, Chinthrajah RS, Chong HJ, Fineman SM, Fleischer DM, Gonzalez-Reyes E, Kim EH, Lanser BJ, MacGinnitie A, Mehta H, Petroni D, Rupp N, Schneider LC, Scurlock AM, Sher LD, Shreffler WG, Sindher SB, Wood R, Yang WH, Sampson HA, Bois T, Green TD, Campbell DE, Bee KJ, Begin P. Long-Term Safety of Epicutaneous Immunotherapy in Peanut-Allergic Children: An Open-Label Active Treatment (REALISE Study). J Allergy Clin Immunol Pract. 2025 May;13(5):1190-1200.e3. doi: 10.1016/j.jaip.2025.02.024. Epub 2025 Feb 27. PMID 40023371